CLINICAL TRIAL: NCT02262286
Title: Study to Procure Human Specimens for Use in the Diagnosis and Management of Traumatic Brain Injury and Other Related Conditions
Brief Title: MIND (Management of Traumatic Brain Injury Diagnosis)
Acronym: MIND
Status: Completed | Type: Observational
Sponsor: Abbott Diagnostics Division (Industry)
Responsible Party: Sponsor
Other Study IDs: 9GP-02-10DELK14
Record Dates: First submitted 2014-09-23; First posted 2014-10-13 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Brain Injury
Keywords: Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples stored at -70C or colder
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Brain Injury: Brain Injury
- Control: Healthy, or Head Trauma, or Orthopedic Trauma, or Poly-Trauma

SUMMARY:
Procure blood specimens from individuals presenting to the emergency department with suspected brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Form Signed
* 18 years of age or older
* For women of child-bearing age: Not known to be pregnant AND
* Head Trauma within 6 hours of ED presentation with Glasgow Coma Scores from 3-8 (Severe Injury), 9-13 (Moderate Injury), or 14-15 (Mild Injury); OR
* Head trauma within 6 hours of ED presentation with Glasgow Coma Score of 15; OR
* Bone fracture or poly-traumas, both with no head trauma

Exclusion Criteria:

* Known pre-existing neurological condition that causes observed symptoms
* Recent history of head injury or seizures (within 1 year of current ED presentation)
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals presenting to the ED within 6 hours of experiencing a head trauma, or bone fractions only.
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Measurement of specific biomarker(s) for brain injury | 48 hours
  Measurement of specific biomarkers to detect brain injury (mild to severe). using 2 or more serial draws from subjects. The biomarkers tested will include established biomarkers s100B, GFAP (Glial Fibrillary Acidic Protein) and also proprietary novel protein and lipid biomarkers that are being studied in discovery research.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Biberthaler, MD/PHD, Principal Investigator — Klinikum reichs der Isar
Locations (1):
- Klinikum rechts der Isar, Munich, Germany